CLINICAL TRIAL: NCT01432977
Title: Paracetamol and Setrons : Drug Interactions in the Management of Pain After Tonsillectomy in Children
Brief Title: Drug Interactions Between Paracetamol and Setrons in Pain Management
Acronym: PARATRON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I10 005
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Droperidol; Ondansetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- comparateur (Active Comparator): paracetamol / droperidol
  Interventions: Drug: paracetamol /droperidol
- Eperimental (Experimental): paracetamol / ondansetron
  Interventions: Drug: paracetamol / ondansetron

INTERVENTIONS:
Drug: paracetamol /droperidol
  Arms: comparateur
Drug: paracetamol / ondansetron
  Arms: Eperimental

SUMMARY:
The aim of this study is to demonstrate that the association paracetamol / ondansetron is not as effective as the association paracetamol / droperidol in the treatment of pain in children following tonsillectomy. The secondary objectives are to compare opioid consumption (morphine / codeine) and the cumulated incidence of nausea and vomiting between the two groups of patients in the first 24 hours after

DETAILED DESCRIPTION:
Tonsillectomy is a common operation performed in children that is associated with marked pain and a high incidence of nausea and vomiting. Therefore, national and international guidelines have recommended the use of a setron as a prevention to nausea and vomiting and also the systematic administration of paracetamol to help in the control of postoperative pain. However, a potential interaction between setrons and paracetamol has been reported in different animal studies and in human volunteers although its existence has never been found in the clinic. Indeed, several hypotheses are proposed to explain the mechanism of action of paracetamol in the treatment of pain. However, a recent one involves the endocannabinoid system and spinal serotonin receptors. Serotonin receptors are also involved in the mechanism of action of antiemetics such as setrons. Indeed, these drugs are serotonin antagonists. Therefore, the investigators hypothesized that the concomitant administration of paracetamol and ondansetron leads to an interaction that will decrease the analgesic effect of paracetamol.

Patients aged 2-7 years old and scheduled for a tonsillectomy will be recruited. They will all receive intraoperatively intravenous paracetamol together with either ondansetron or droperidol. Pain scores using the CHEOPS scale will be recorded for 24 hours. Furthermore, patients will receive i.v. morphine during the operation and in the recovery room if necessary and a non-steroidal anti-inflammatory drug for postoperative pain; on the ward, oral codeine will be administered when needed. Pain scores will be recorded regularly for up to 24 hours together with opioid consumption and the incidence of nausea and vomiting in the same period. Any adverse event will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* tonsillectomy in a child 2-7 years old who is hospitalized for at least 24 hours ;
* informed consent from one parent at least

Exclusion Criteria:

* hospital stay of less than 24 hours ;
* patient already on pain medication ;
* allergic patient with a contra-indication to one of the study drugs.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
-pain scores | 4 hours after drug administration
  pain scores at rest 4 hours after administration of paracetamol and ondansetron / droperidol intraoperatively

SECONDARY OUTCOMES:
analgesic consumption | 24 hours after inclusion
  analgesic consumption during 24 hours podt inclusion
incidence of nausea and vomiting. | data continuiousley collected during 24 hours
  - incidence of nausea and vomiting.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chirurgie Ped, Limoges
  - Service Anesthésie, Limoges